CLINICAL TRIAL: NCT00075881
Title: Phase II Study of PS-341 for Patients With High-Risk, Newly Diagnosed Multiple Myeloma
Brief Title: Bortezomib in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00652; NCI-2014-00652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000349450; E2A02 (Other: Eastern Cooperative Oncology Group); E2A02 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-03

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bortezomib) (Experimental): INDUCTION TREATMENT: Patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE TREATMENT: Patients who complete induction treatment without progressive disease receive bortezomib IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  REINDUCTION TREATMENT: Patients who progress while on maintenance treatment receive bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial studies how well bortezomib works in treating patients with newly diagnosed multiple myeloma. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate to PS-341 (bortezomib) induction in patients with high risk, newly diagnosed multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate progression free survival. II. To explore the response rate of patients who relapse or progress on maintenance and then return to induction schedule.

III. To explore duration of second response.

TERTIARY OBJECTIVES:

I. To explore a possible differential response to PS-341 with previously described adverse prognostic indicators.

II. To explore specific gene expression profiles (GEP) that may predict response to therapy to an agent or combination of agents used in the treatment of newly diagnosed myeloma.

III. To explore specific post-treatment gene expression profiles (GEP) in the patients who have received 4 cycles of therapy and achieved a minimal response or better.

IV. To develop relevant information about the immune system for multiple myeloma patients treated with PS-341.

OUTLINE:

INDUCTION TREATMENT: Patients receive bortezomib intravenously (IV) on days 1, 4, 8, and 11. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE TREATMENT: Patients who complete induction treatment without progressive disease receive bortezomib IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

REINDUCTION TREATMENT: Patients who progress while on maintenance treatment receive bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must not have received prior myeloma specific therapy (chemotherapy, radiotherapy, or biologic therapy) other than bisphosphonate therapy

  * Patients may have received radiation of plasmacytoma (for example, solitary plasmacytoma); the last such treatment must have occurred >= 4 weeks prior to registration
* Patients must be recently diagnosed with symptomatic multiple myeloma confirmed by meeting one or more of the following criteria (obtained =< 30 days prior to registration):

  * NOTE: serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP) and marrow biopsy all must be done at baseline in order to evaluate response

    * Monoclonal protein in the serum >= 1 g/dl (measurable disease), or
    * Monoclonal light chain in the urine protein electrophoresis >= 200 mg/24 hours (measurable disease), or
    * Bone marrow plasmacytosis >= 30% without either of the values in above (evaluable disease)
* Patients must meet one or more of the following (all tests must be been drawn =< 30 days prior to registration but all results are not required to be available at time of registration as long as at least one of the following criteria has been met; if patient is otherwise eligible, plasma cell labeling index [PCLI] is not required, but is requested):

  * Beta-2 microglobulin >= 5.5 mcg/mL, or
  * PCLI >= 1, or
  * Deletion 13 by cytogenetics
* Platelet count >= 20,000/mm^3, with or without transfusion support
* Hemoglobin >= 7.0 g/dL, with or without transfusion support
* Absolute neutrophil count (ANC) >= 500/mm^3 without growth factor support
* Direct bilirubin within =< 1.5 x upper normal limits (UNL)
* Alkaline phosphatase =< 2.5 x UNL
* Aspartate aminotransferase (AST) =< 2.5 x UNL
* Calculated or measured creatinine clearance >= 20 mL/minute
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2; exception: PS = 3 if secondary to acute bone event (fracture)
* Patients may not receive concurrent chemotherapy, radiotherapy or biologic therapy while on study; the exception for corticosteroids is made for those taking chronic corticosteroids for disorders other than myeloma, such as rheumatoid arthritis, adrenal insufficiency, etc.

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Patients must not have a history of allergic reaction attributable to compounds containing boron or mannitol
* Patient must not have a peripheral neuropathy > grade 1, as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 3.0):

  * Grade 2: Objective sensory (or motor) loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living (ADL)
  * Grade 3: Sensory (or motor) loss or paresthesia interfering with ADL
  * Grade 4: Permanent sensory (or motor) loss that interferes with function
* Patient must be capable of understanding the investigational nature, potential risks and benefits of the study
* Patient must have adequate cardiac function; patient must not have:

  * History of a myocardial infarction within 6 months of enrollment
  * New York Heart Association (NYHA) class III or IV heart failure
  * Uncontrolled angina or electrocardiographic evidence of acute ischemia
  * Severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of active conduction system abnormalities
  * Cardiac amyloidosis
* Patient must not have any other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Patient must not have poorly controlled hypertension
* Women must not be pregnant or breast feeding; all females of childbearing potential must have a blood test or urine study within 7 days prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on January 16, 2004 and terminated on March 7, 2005 after 44 patients had enrolled. Accrual rate was 3 patients per month, slower than expected rate (6 patients per month)
Groups:
- PS-341: Induction treatment: PS-341 1.3 mg/m2 IV push days 1, 4, 8, and 11. As per the PS-341 package insert, there should be at least 72 hours between each PS-341 dose. Repeat cycles every 3 weeks for a total of 8 cycles.
  Maintenance treatment: PS-341 1.3 mg/m2 IV push days 1 and 15.
  Reinduction treatment: PS-341 1.3 mg/m2 IV push days 1, 4, 8, and 11. As per the PS-341 package insert, there should be at least 72 hours between each PS-341 dose.
Period: Overall Study
Arm/Group | PS-341
Started | 44
Eligible | 43
Treated | 42
Induction Treatment | 42
Maintenance Treatment | 15
Reinduction Treatment | 7
Completed | 1
Not Completed | 43
Not completed — Lack of Efficacy | 18
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 4
Not completed — other complicating disease | 3
Not completed — other | 4
Not completed — missing data | 2
Not completed — Ineligible | 1
Not completed — never start protocol therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | PS-341
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 63 [44 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate on Induction
Description: Eastern Cooperative Oncology Group (ECOG) Myeloma Response Criteria that follows the standard European Group for Blood and Bone Marrow Transplant criteria was used to evaluate patient response and progression. Patients who have complete disappearance of an M-protein and no evidence of myeloma in the bone marrow are considered to have complete response. 42 eligible and treated patients were included in the analysis.
Time Frame: participants were evaluated prior to each cycle, up to 8 cycles with a median number of 6 cycles. 1 cycle=21 days
Population: 42 eligible and treated patients were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- PS-341: Induction treatment: PS-341 1.3 mg/m2 IV push days 1, 4, 8, and 11. As per the PS-341 package insert, there should be at least 72 hours between each PS-341 dose. Repeat cycles every 3 weeks for a total of 8 cycles.
  Maintenance treatment: PS-341 1.3 mg/m2 IV push days 1 and 15
  Reinduction treatment: PS-341 1.3 mg/m2 IV push days 1, 4, 8, and 11. As per the PS-341 package insert, there should be at least 72 hours between each PS-341 dose.
Arm/Group | PS-341
Number analyzed (Participants) | 42
percentage of participants | 47.6 [34.2 to 61.3]

2. Secondary Outcome: Response Rate on Maintenance
Description: ECOG Myeloma Response Criteria that follows the standard European Group for Blood and Bone Marrow Transplant criteria was used to evaluate patient response and progression. Patients who have complete disappearance of an M-protein and no evidence of myeloma in the bone marrow are considered to have complete response. 15 eligible and treated patients were included in the analysis.
Time Frame: participants were evaluated prior to each cycle, up to 45 cycles with a median number of 9 cycles. 1 cycle=21 days
Population: 15 eligible and treated patients were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- PS-341: Maintenance treatment: PS-341 1.3 mg/m2 IV push days 1 and 15
Arm/Group | PS-341
Number analyzed (Participants) | 15
percentage of participants | 66.7 [42.3 to 85.8]

3. Secondary Outcome: Response Rate on Reinduction
Description: ECOG Myeloma Response Criteria that follows the standard European Group for Blood and Bone Marrow Transplant criteria was used to evaluate patient response and progression. Patients who have complete disappearance of an M-protein and no evidence of myeloma in the bone marrow are considered to have complete response. 7 eligible and treated patients were included in the analysis.
Time Frame: participants were evaluated prior to each cycle, up to 23 cycles with a median number of 3 cycles. 1 cycle=21 days
Population: 7 eligible and treated patients were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- PS-341: Reinduction treatment: PS-341 1.3 mg/m2 IV push days 1, 4, 8, and 11. As per the PS-341 package insert, there should be at least 72 hours between each PS-341 dose
Arm/Group | PS-341
Number analyzed (Participants) | 7
percentage of participants | 28.6 [5.4 to 65.9]

4. Secondary Outcome: 1-year Progression Free Survival Probability
Description: Progression-free survival is defined as time from randomization to disease progression or death from any cause, whichever occurred first. Disease progression is defined using the ECOG Myeloma Response Criteria. Kaplan-Meier method is used to estimate the 1-year progression-free survival probability. 42 eligible and treated patients were included in the analysis.
Time Frame: Every 3 months if patient is <2 years from study entry, every 6 months if patient is 2-6 years from study entry, no specific requirment if patient is more than 6 years from study entry
Population: 42 eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PS-341
Number analyzed (Participants) | 42
percentage of participants | 36.4 [19.4 to 53.7]

ADVERSE EVENTS:
Time Frame: Reported at the end of each cycle on treatment and at 30 days following the last dose of treatment. Reported every 3 months within 2 years of study entry, and every 6 months between 2-6 years of study entry
Description: 1 cycle = 21 days for induction and re-induction, 1 cycle=28 days for maintenance
Arm/Group | PS-341
Serious Adverse Events (participants affected / at risk) | 37/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PS-341 (N=43)
Anemia (Blood and lymphatic system disorders) | 12
Leukopenia (Investigations) | 9
Neutropenia (Investigations) | 14
Thrombocytopenia (Investigations) | 8
Heart block asystole (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Vasovagal episode (Nervous system disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Fatigue (General disorders) | 7
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 2
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Edema limb (General disorders) | 1
Alkaline phosphatase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Boold amylase increased (Investigations) | 1
Aspartate aminotransferase (AST) increased (Investigations) | 1
Bilirubin increased (Investigations) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3
Creatinine increased (Investigations) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 9
Confusion (Psychiatric disorders) | 1
Dizziness/lightheadedness (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Abonominal pain (Gastrointestinal disorders) | 3
Muscle pain (Musculoskeletal and connective tissue disorders) | 2
Neuropathic pain (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PS-341 (N=43)
Anemia (Blood and lymphatic system disorders) | 38
Leukopenia (Investigations) | 27
Neutropenia (Investigations) | 27
Thrombocytopenia (Investigations) | 31
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 6
Fatigue (General disorders) | 29
Fever w/o neutropenia (General disorders) | 6
Weight loss (Investigations) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 22
Constipation (Gastrointestinal disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 14
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 26
Taste disturbance (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Edema limb (General disorders) | 6
Alkaline phosphatase increased (Investigations) | 17
Alanine aminotransferase (ALT) increased (Investigations) | 11
Aspartate aminotransferase (AST) increased (Investigations) | 15
Bilirubin increased (Investigations) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 23
Creatinine increased (Investigations) | 19
Hyperkalemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypernatremia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 20
Dizziness/lightheadedness (Nervous system disorders) | 12
Neuropathy-motor (Nervous system disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 25
Abonominal pain (Gastrointestinal disorders) | 8
Headache (Nervous system disorders) | 3
Join pain (Musculoskeletal and connective tissue disorders) | 10
Muscle pain (Musculoskeletal and connective tissue disorders) | 11
Neuropathic pain (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less